CLINICAL TRIAL: NCT06927687
Title: A Phase II Study to Evaluate Efficacy, Safety, and Pharmacokinetics of ZG005 in Patients With Advanced Solid Tumors
Brief Title: Study of ZG005 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZG005-001-02
Record Dates: First submitted 2025-04-07; First posted 2025-04-15 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose Expansion (Experimental): ZG005 dose expansion was performed in different tumors, such as: nasopharyngeal carcinoma, esophageal squamous cell carcinoma, and other carcinoma
  Interventions: Biological: ZG005 for Injection

INTERVENTIONS:
Biological: ZG005 for Injection — Recommended Phase 2 Dose (RP2D) of ZG005(20 mg/kg), intravenous infusion, once every 3 weeks.
  Other Names: ZG005

SUMMARY:
This is an open-label, multicenter, Phase II clinical trial, designed to evaluate the efficacy and safety of ZG005 in patients with advanced solid tumors who have previously failed or are intolerant to standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* Fully understand the study and voluntarily sign the informed consent form.
* Male or female 18-75 years of age;
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1;
* Life expectancy ≥ 12 weeks;
* Histologically or cytologically confirmed diagnosis of advanced solid tumors.

Exclusion Criteria:

* Medical history, computed tomography (CT) or magnetic resonance imaging (MRI) results indicate that existence of the central nervous system(CNS) metastases;
* Any other malignancy within 5 years.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-13 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Objective response rate(ORR) | Up to 2 years

SECONDARY OUTCOMES:
Adverse Event (AE) | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jason Wu, Study Chair — Suzhou Zelgen Biopharmaceuticals Co.,Ltd
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China